CLINICAL TRIAL: NCT00067730
Title: A Safety Evaluation of Xigris Drotrecogin Alfa Activated in Hematopoietic Stem Cell Transplant Patients With Severe Sepsis
Brief Title: A Safety Evaluation of Drotrecogin Alfa (Activated) in Patients With Blood Cancer, Severe Infection Related to Bone Marrow Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6416; F1K-US-EVCE
Record Dates: First submitted 2003-08-25; First posted 2003-08-27 (Estimated); Last update posted 2007-12-07 (Estimated); Status verified 2007-12

CONDITIONS: Sepsis; Hematologic Neoplasms; Hematopoietic Stem Cell Transplantation; Infection
MeSH Terms: conditions — Sepsis; Hematologic Neoplasms; Infections | interventions — drotrecogin alfa activated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 24 microgram/kg/hr for 96 hours (+ or - 1 hour)
  Interventions: Drug: Drotrecogin Alfa (activated)

INTERVENTIONS:
Drug: Drotrecogin Alfa (activated)
  Other Names: LY203638; Xigris

SUMMARY:
The purpose is to determine how Drotrecogin Alfa (activated) will affect patients with blood cancers who develop severe sepsis within 60 days of starting chemotherapy in preparation for bone marrow transplant (BMT).

DETAILED DESCRIPTION:
The purpose of this study is to determine how Drotrecogin Alfa (activated) will affect leukemia, lymphoma and myeloma patients who develop sever sepsis within 60 days of starting chemotherapy in preparation for bone marrow transplant (BMT). The study will evaluate the safety of Xigris by assessing the risk of serious bleeding events, including bleeding within the brain and serious bleeding leading to death.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have Leukemia, Lymphoma or Myeloma.
* Participants must have had hematopoietic stem cell transplantation(HSCT) within the past 60 days.
* Participants must have infection with either vasopressor dependent septic shock or ventilator-dependent respiratory failure.
* Participants must be on a breathing machine or require medication to maintain their blood pressure.

Exclusion Criteria:

* Participants must not have increased bleeding risk due to medical conditions or medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2003-03; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Safety | 10 months

SECONDARY OUTCOMES:
Mortality | 10 months
Bleeding incidence | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iowa City, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manhassaet, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winston-Salem, North Carolina

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com